CLINICAL TRIAL: NCT05728827
Title: Rehabilitation With Blood Flow Restriction Training to Enhance Anti-gravity Treadmill Effects in the Treatment of Patients With Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: A Study to Compare Two Rehabilitation Protocols for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-39
Record Dates: First submitted 2023-02-03; First posted 2023-02-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-gravity treadmill + Blood Flow Restriction training (Experimental)
  Interventions: Other: Blood flow restriction training + Anti-gravity treadmill
- Anti-gravity treadmill (Active Comparator)
  Interventions: Other: Anti-gravity treadmill

INTERVENTIONS:
Other: Blood flow restriction training + Anti-gravity treadmill — Blood flow restriction training is administered via straps applied to the proximal limb with the possibility to adjust the applied occlusion pressure in order to prevent venous return leaving the arterial flow partially free. The consequent blood pooling causes a reduction in tissue saturation with oxidative stress and an increased growth factors secretion. The intervention will be applied while walking/running on the anti-gravity treadmill.
  Arms: Anti-gravity treadmill + Blood Flow Restriction training
Other: Anti-gravity treadmill — The intervention will be applied walking/running on the anti-gravity treadmill.
  Arms: Anti-gravity treadmill

SUMMARY:
The aim of this randomized controlled study is to investigate whether the implementation of Blood Flow Restriction, in which the de-loading factor is delivered by the combined progressive de-loaded walking to running activity on an antigravity treadmill (treatment group), is more effective than the same antigravity protocol alone (control group).

Participants will be divided as follows:

Intervention group: anti-gravity treadmill combined with blood flow restriction Control group: anti-gravity treadmill Both groups will also undergo a standardized knee Osteoarthritis management through an aerobic and strength program.

ELIGIBILITY:
Inclusion Criteria:

* Age included between 45 and 80 years old
* Patients with knee OA diagnosed by a medical doctor with a radiological confirmation
* Patients able to provide informed consent and follow all the study procedures as indicated by the protocol
* Informed Consent as documented by signature

Exclusion Criteria:

* Younger than 44 years old or older than 81 years old included
* Known drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another study with an investigational drug within the 30 days preceding and during the present study
* Treatment with an injective approach in the previous 3 month
* Surgical treatment in the previous 12 months.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Post-operative knee outcome on Western Ontario and McMaster Universities Arthritis Index | Change from Baseline to 6 months
  Questionnaire at baseline (day 1) and 6 weeks, and at 3, 6 months. The WOMAC questionnaire is composed of 3 sub-scores that evaluate pain (5 questions, 0-20 points), stiffness (2 questions, 0-8 points), and function (17 questions, 0-68 points) and is a validated patient-reported outcome measure (PROM) to evaluate knee osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, MD, Study Chair — EOC
Locations (1):
- Christian Candrian, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No